CLINICAL TRIAL: NCT06049485
Title: Unveiling Follicular Lymphoma Clinical Trials: Analyzing Patient Engagement Patterns and Participation Trends
Brief Title: Assessing the Experience of Patients Undergoing Follicular Lymphoma Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 70732724
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, participation in medical studies is highly skewed towards particular demographic groups of people.

This research will invite several participants to gather a wide range of information on clinical trial experiences for follicular lymphoma patients. The aim of the study is to identify the factors that limit the ability of a person to enroll in, as well as complete a clinical trial for treatment of follicular lymphoma.

The data collected from this study will help improve future outcomes for all follicular lymphoma patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age or older
* Patient has been diagnosed with follicular lymphoma
* Patient has access to a home internet connection in order to provide regular updates through the course of the study

Exclusion Criteria:

* Women of childbearing potential without a negative pregnancy test; or women who are lactating.
* Inability to provide written informed consent
* Patients receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with follicular lymphoma who are actively considering enrolling in a medical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a follicular lymphoma clinical research | 3 months
Rate of patients who remain in a follicular lymphoma medical study to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gueiderikh A, Ung M, Lazarovici J, Danu A, Ghez D, Saleh K, Dragani M, Noel N, Bigenwald C, Willekens C, Ribrag V, Michot JM, Martin V. Incidence, characteristics, management and outcome of patients with follicular lymphoma with tumor epidural compression, a study on 22 cases. Cancer Radiother. 2023 Sep;27(5):370-375. doi: 10.1016/j.canrad.2023.04.004. Epub 2023 May 6. PMID 37156711
- [Background] Friedberg JW, Taylor MD, Cerhan JR, Flowers CR, Dillon H, Farber CM, Rogers ES, Hainsworth JD, Wong EK, Vose JM, Zelenetz AD, Link BK. Follicular lymphoma in the United States: first report of the national LymphoCare study. J Clin Oncol. 2009 Mar 10;27(8):1202-8. doi: 10.1200/JCO.2008.18.1495. Epub 2009 Feb 9. PMID 19204203
- [Background] Ruella M, Filippi AR, Bruna R, Di Russo A, Magni M, Caracciolo D, Passera R, Matteucci P, Di Nicola M, Corradini P, Parvis G, Gini G, Olivieri A, Ladetto M, Ricardi U, Tarella C, Devizzi L. Addition of Rituximab to Involved-Field Radiation Therapy Prolongs Progression-free Survival in Stage I-II Follicular Lymphoma: Results of a Multicenter Study. Int J Radiat Oncol Biol Phys. 2016 Mar 15;94(4):783-91. doi: 10.1016/j.ijrobp.2015.12.019. Epub 2015 Dec 17. PMID 26972651

DOCUMENTS (1):
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT06049485/ICF_000.pdf